CLINICAL TRIAL: NCT00560898
Title: Comparison of Two Multi-Purpose Solution and Contact Lens Material Combinations on Human Corneal Barrier Function
Brief Title: Comparison of Two Multi-Purpose Solution and Lens Material Combinations on Corneal Barrier Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Collaborators: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 00001418; 00001418
Record Dates: First submitted 2007-11-15; First posted 2007-11-20 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Contact Lens Disinfecting Solutions
Keywords: staining; epithelial barrier function

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 (Experimental): contact lenses disinfected in multipurpose solution
  Interventions: Drug: ProClear Lens Material soaked in ReNu Multiplus Multipurpose Solution
- 3 (Experimental): contact lenses disinfected in multipurpose solution
  Interventions: Drug: Acuvue Advance Lens Material soaked in ReNu Multiplus Multipurpose Solution
- 4 (Experimental): contact lenses disinfected in multipurpose solution
  Interventions: Drug: Acuvue Advance Lens Material soaked in Optifree RepleniSH Multipurpose Solution
- 1 (Experimental): contact lenses disinfected in multipurpose solution
  Interventions: Drug: ProClear Lens Material soaked in Optifree RepleniSH Multipurpose Solution

INTERVENTIONS:
Drug: ProClear Lens Material soaked in ReNu Multiplus Multipurpose Solution — Contact lens soaked in multipuprpose solution for 8 hours, then worn for two hours
  Arms: 2
Drug: Acuvue Advance Lens Material soaked in ReNu Multiplus Multipurpose Solution — Contact lens soaked in multipuprpose solution for 8 hours, then worn for two hours
  Arms: 3
Drug: Acuvue Advance Lens Material soaked in Optifree RepleniSH Multipurpose Solution — Contact lens soaked in multipuprpose solution for 8 hours, then worn for two hours
  Arms: 4
Drug: ProClear Lens Material soaked in Optifree RepleniSH Multipurpose Solution — Contact lens soaked in multipuprpose solution for 8 hours, then worn for two hours
  Arms: 1

SUMMARY:
The purpose of this study is to measure the relative "barrier" function of the top layer of the cornea (called the epithelium), or the degree to which the cornea can prevent the penetration of the colored dye sodium fluorescein into the eye. This is a clinical investigation of the effect on corneal barrier function following wear of two contact lens materials and two contact lens care systems, approved for marketing in the US by the Food and Drug Administration. These contact lenses will be worn for two hours, following soak in one of two marketed contact lens disinfecting solutions. Approximately 25 young, adapted contact lens wearers will participate.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.

  * Understand your rights as a research subject and give written informed consent by signing the Informed Consent Form, Subject Bill of Rights, and Patient Authorization for Use and Release of Health and Research Study Information (HIPAA form).
  * Be likely to finish the entire study, understand the study instructions, and be willing to follow the instructions.
  * Contact lens prescription between +4.00 D to -9.00 D (spherical equivalent).
  * Best correctable visual acuity of at least 20/40 in each eye.
  * Willing to de-adapt (do not wear) from habitual contact lenses for periods of three days prior to barrier function determination.
  * Possess a functional spectacle prescription to allow adequate vision during the de-adaptation and barrier function determination periods.
  * No known ocular or systemic allergies, which may interfere with contact lens wear.
  * No known systemic disease, or need for medication that may interfere with contact lens wear (i.e. antihistamines, beta-blockers, steroids).

Exclusion Criteria:

* Subjects demonstrating any medical condition that may affect the results of this study SHOULD NOT be enrolled. The following are specific conditions that exclude subjects from enrollment in this study.

  * Eye (ocular) or systemic allergies that may interfere with contact lens wear.
  * Less than one month successful, full time (defined as more than 8 hours per day, and more than 5 days per week) soft lens wear.
  * Systemic disease or uses of medication, which may interfere with contact lens wear.
  * Clinically significant corneal swelling (greater than grade 3 or 4 on a 0-4 scale), corneal blood vessel growth) (vascularization), corneal staining, bulbar redness, tarsal redness, or any other abnormality of the cornea that may cause unsafe contact lens wear.
  * Any active ocular infection.
  * Prior corneal refractive surgery (i.e., LASIK, PRK, etc).
  * Have used medications within 24 hours of study entry or have an ongoing need to use ocular medication.
  * Are taking part in any other study or have taken part in a study within the last 14 days
  * Have a medical condition that your study eye doctor thinks may make it not appropriate for you to participate in this study.
  * Are pregnant, or anticipate becoming pregnant during the course of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Epithelial penetration rate of sodium fluoeescein, in nm/sec | Immediately post measurement

SECONDARY OUTCOMES:
Corneal staining | Immediately following barrier determination

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Paugh, OD, PhD, Principal Investigator — Southern California College of Optometry at Marshall B. Ketchum University
Locations (1):
- Southern California College of Optometry, Fullerton, California, United States